CLINICAL TRIAL: NCT00523445
Title: Varenicline, an Alpha 4 Beta 2 Nicotinic Acetylcholine Receptor Partial Agonist, on Cognitive Dysfunction in 120 Patients With Schizophrenia: a Randomized, Double Blind, 8 Weeks Trial
Brief Title: The Effects of Varenicline on Cognitive Function in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inje University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Joo Shim, Inje University Busan Paik Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Varenicline07; 07TAS-1051
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognition; Varenicline
MeSH Terms: conditions — Schizophrenia | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): The effect of varenicline on cognitive function of Varenicline(Chantix) is being compared to that of placebo
  Interventions: Drug: Varenicline(Chantix)
- Placebo (Placebo Comparator): The effect of placebo comparator is being compared to that of varenicline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline(Chantix) — The dose of antipsychotic drug will remain fixed throughout the study and the titration of varenicline will be as follows: varenicline 0.5 mg/d for days 1 to 3, 0.5 mg twice per day for days 4 to 7, then 1 mg twice per day through week 8.
  Arms: Varenicline
Drug: Placebo — The dose of antipsychotic and concomitant medications remained fixed throughout the study and the titration of varenicline was as follows: Placebo will be supplied twice daily through week 8.
  Arms: Placebo

SUMMARY:
The primary objective of this project is to examine the effects of varenicline treatment used concomitantly with antipsychotic medications, on cognitive dysfunction in people with schizophrenia. The secondary objective is to evaluate the effect of this combination therapy on smoking in people with schizophrenia. This study will be a randomized, double blind, parallel group, placebo controlled 8 weeks trial.

DETAILED DESCRIPTION:
Cognitive deficits have been considered as a core symptom domain of schizophrenia. Amelioration of or improvement in cognitive impairments is becoming an important focus of clinical treatment development. Varenicline is a potent and selective alpha 4 beta 2 nicotinic acetylcholine receptor partial agonist that has been developed for smoking cessation. In animal studies, alpha 4 beta 2 receptor agonists significantly improve working memory and attention function. Subjects will be assigned in 1:1 ratio to receive varenicline or placebo respectively. Assessments will be done using several neuropsychologic tests, clinical rating scale including assessment of nicotine withdrawal scales.Varenicline has been found to be efficacious for smoking cessation in the general population and animal studies have demonstrated the cognitive benefits of this agent. However, no published work is available evaluating the cognitive effects in humans. Thus, patients may experience improvements in cognitive function and in people who are smokers, these people may be able to achieve abstinence in smoking. This will in turn improve long-term functional outcomes and health outcomes in people with schizophrenia. This is an exciting opportunity for discovery if indeed cognitive abilities could be improved with this adjunctive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients with schizophrenia

Exclusion Criteria:

* Refractory schizophrenia
* Mental Retardation
* Serious Medical illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To examine the effects of varenicline treatment used concomitantly with antipsychotic medications, on cognitive dysfunction in people with schizophrenia. | 8 weeks

SECONDARY OUTCOMES:
To evaluate the effect of this combination therapy on smoking in people with schizophrenia. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Cheol Shim, MD.PhD, Principal Investigator — Inje University
Locations (5):
- South Korea (5):
  - Dongrae Hospital, Busan
  - Jamyeong, Busan
  - Busan Paik Hospital, Busan
  - Ahab Hospital, Busan
  - Dongseo hospital, Masan

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Jeon DW, Shim JC, Kong BG, Moon JJ, Seo YS, Kim SJ, Oh MK, Jung DU. Adjunctive varenicline treatment for smoking reduction in patients with schizophrenia: A randomized double-blind placebo-controlled trial. Schizophr Res. 2016 Oct;176(2-3):206-211. doi: 10.1016/j.schres.2016.08.016. Epub 2016 Aug 16. PMID 27543252
- [Derived] Shim JC, Jung DU, Jung SS, Seo YS, Cho DM, Lee JH, Lee SW, Kong BG, Kang JW, Oh MK, Kim SD, McMahon RP, Kelly DL. Adjunctive varenicline treatment with antipsychotic medications for cognitive impairments in people with schizophrenia: a randomized double-blind placebo-controlled trial. Neuropsychopharmacology. 2012 Feb;37(3):660-8. doi: 10.1038/npp.2011.238. Epub 2011 Nov 2. PMID 22048460